CLINICAL TRIAL: NCT03988322
Title: Computed Tomography Screening for Early Lung Cancer, COPD and Cardiovascular Disease in Shanghai: a Population-based Comparative Study
Brief Title: Computed Tomography Screening for Early Lung Cancer, COPD and Cardiovascular Disease in Shanghai, China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Liu ShiYuan, Professor, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016YFE0103000
Record Dates: First submitted 2019-06-07; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Lung Neoplasms; Mass Screening; Chronic Obstructive Pulmonary Disease; Cardiovascular Disease
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quantitative assessment of imaging biomarkers (Experimental): This is the intervention arm. In this arm, the participants will be scanned with low-dose CT with pre-defined scanning parameters for two rounds (at baseline and in the second year). The screen-detected lung nodules will be managed according to the volume of the nodule. The quantitative assessment of imaging biomarkers of lung cancer, COPD and cardiovascular disease will be recorded.
  Interventions: Other: Low-dose CT screening with quantitative assessment and management of imaging biomarkers
- Visual assessment of imaging biomarkers (Active Comparator): This is the control arm. In this arm, the participants will be scanned with low-dose CT with routine scanning parameters used for lung cancer screening in the hospital for two rounds (at baseline and in the second year). The screen-detected lung nodules will be managed according to the diameter of the nodule. The imaging biomarkers related to lung cancer, COPD and cardiovascular disease will be visually assessed.
  Interventions: Other: Low-dose CT screening with visual assessment and management of imaging biomarkers

INTERVENTIONS:
Other: Low-dose CT screening with quantitative assessment and management of imaging biomarkers — Participants will be screened with a low-dose CT (a Philips 256-slice CT system). The CT images will be obtain according to the pre-defined CT scan protocol. This CT protocol is developed for quantitative assessment of lung nodules, COPD and coronary artery calcium. Detected lung nodules will be managed according to the European volume-based protocol, based on the volume and volume doubling time of lung nodule. COPD will be management according to the result of lung function test. The imaging biomarkers (eg., emphysema index, airway wall thickness, and coronary artery calcium ) will be quantitatively registered. In addition, a number of participants' characteristics will be collected: physical examination (weight, height, blood pressure), laboratory measurements (eg., fasting plasma glucose, total cholesterol, HDL-cholesterol). The social-demographic characteristics, risk factors of the 3 diseases, and health status of the participants will be collected through questionnaires.
  Arms: Quantitative assessment of imaging biomarkers
Other: Low-dose CT screening with visual assessment and management of imaging biomarkers — Participants will be screened with a low-dose CT (a Philips 64 MDCT system). The CT images will be obtain according to the routine CT scan protocol for lung cancer screening in the hospital. Detected lung nodules will be managed according to the diameter of the nodule based on the NCCN Clinical Practice Guideline in Oncology for Lung Cancer Screening. Detected emphysema and/or bronchial wall thickness, coronary artery calcium will be qualitatively recorded (yes/no).
  Arms: Visual assessment of imaging biomarkers

SUMMARY:
Low-dose chest computed tomography (CT) is considered as a screening method for early detection of lung cancer in the population at risk, and it also allows to detect chronic obstructive pulmonary disease (COPD) and cardiovascular disease (CVD). Studies in European population showed the benefit of volumetric assessment of CT screening-detected lung nodules compared to diameter-based assessment. Screening for COPD and CVD, in addition to lung cancer, may significantly increase the benefits of low-dose CT lung cancer screening. The objective is to assess the screening performance of volume-based management of CT-detected lung nodule in comparison to diameter-based management, and to improve the effectiveness of CT screening for COPD and CVD, in addition to lung cancer, based on quantitative measurement of CT imaging biomarkers in a Chinese screening setting. Thus, a population-based comparative study will be performed in Shanghai, China.

DETAILED DESCRIPTION:
The study will recruit 10,000 asymptomatic participants between 40 and 74 years old from Shanghai urban population. The 5000 participants in the intervention group will undergo a low-dose CT scan at baseline and one year later, and will be managed according to European volume-based protocol. The 5000 participants in the control group will undergo a low-dose CT scan according to the routine CT protocol and will be managed according to the clinical practice. Epidemiological data will be collected through questionnaires. In the fourth year from baseline, the diagnosis of the three diseases will be collected. The screening performance will be compared between volume-based and standard protocol for managing early-detected lung nodules. The effectiveness of quantitative measurement of CT imaging biomarkers for early detection of lung cancer, COPD and CVD will be evaluated.

The detected lung nodules in the intervention group will be classified into three groups depending on nodule volume: < 100 mm3 (negative result), 100-300 mm3 (indeterminate result) and > 300 mm3 (positive result). In case of a negative result, a CT scan after one year is recommended. In case of an indeterminate result, a 3-month follow up CT is recommended at which VDT will be assessed. For short VDT (< 400 days), the screening result is positive. Long VDT (> 400 days) is considered a negative screening result. In case of a positive result, referral to a multidisciplinary team is recommended for further investigation. The detected nodules in the control group will be managed according to the recommended cut-off values of diameter from NCCN Clinical Practice Guideline in Oncology for Lung Cancer Screening.

ELIGIBILITY:
Inclusion Criteria:

1. asymptomatic (without complaints of chest discomfort) residents registered in Shanghai city.
2. age between 40-74 years old
3. no history of lung cancer (self-reported).

Exclusion Criteria:

* Pregnant women will be excluded.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
number of incident lung cancer | at the fourth year from baseline
  The number of clinically diagnosed lung cancer will be collected through the Hospital Information System (HIS) of Shanghai Changzheng Hospital and from the general practitioners by using a pre-defined questionnaire.
number of COPD | at the fourth year from baseline
  The number of clinically diagnosed COPD, the number of hospitalization due to COPD and the number of acute exacerbation will be collected through the Hospital Information System (HIS) of Shanghai Changzheng Hospital and from the general practitioners by using a pre-defined questionnaire.
number of cardiovascular event | at the fourth year from baseline
  The number of cardiovascular event(eg, major adverse cardiovascular event, myocardial infarction, stroke)will be collected through the Hospital Information System (HIS) of Shanghai Changzheng Hospital and from the general practitioners by using a pre-defined questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyuan Liu, Prof, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and publications of study results will be shared.
Supporting Information: Study Protocol
Time Frame: The study protocol will be available from January 2020. The study results will be available when published.
Access Criteria: All sharing will be accessed by publications, national and international scientific conference.

REFERENCES:
- [Derived] Du Y, Li Q, Sidorenkov G, Vonder M, Cai J, de Bock GH, Guan Y, Xia Y, Zhou X, Zhang D, Rook M, Vliegenthart R, Heuvelmans MA, Dorrius MD, van Ooijen PMA, Groen HJM, van der Harst P, Xiao Y, Ye Z, Xie X, Wang W, Oudkerk M, Fan L, Liu S. Computed Tomography Screening for Early Lung Cancer, COPD and Cardiovascular Disease in Shanghai: Rationale and Design of a Population-based Comparative Study. Acad Radiol. 2021 Jan;28(1):36-45. doi: 10.1016/j.acra.2020.01.020. Epub 2020 Mar 6. PMID 32151538